CLINICAL TRIAL: NCT06879665
Title: TANDem-2: Closing the Gap to Interventions for TAND
Acronym: TANDem-2
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: University of Cape Town (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Prof Anna Jansen, Professor, Vrije Universiteit Brussel
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-2024-222; HT94252410790 (Other Grant/Funding Number: US Department of Defense); HT94252410791 (Other Grant/Funding Number: US Department of Defense); 327/2024 (Other Grant/Funding Number: University of Cape Town Human Research Ethics Committee)
Record Dates: First submitted 2025-02-28; First posted 2025-03-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Adult Caregivers of Individuals With TSC; Tuberous Sclerosis Complex (TSC)
Keywords: Caregiver well-being; Psychological flexibility; Acceptance and Commitment Therapy (ACT); Tuberous sclerosis complex (TSC); TSC-Associated Neuropsychiatric Disorders (TAND)
MeSH Terms: conditions — Tuberous Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Feasibility of "Well-Beans for Caregivers" (Other): Pre-post- quazi-experimental pilot intervention of the feasibility, acceptability and impact of the "Well-Beans for Caregivers" Program
  Interventions: Behavioral: Well-Beans for Caregivers Program

INTERVENTIONS:
Behavioral: Well-Beans for Caregivers Program — This is a brief behavioral intervention consisting of 3 weekly 2-hour sessions. The sessions are based on Acceptance and Commitment Therapy (ACT) and are designed to improve psychological flexibility in caregivers. This in turn is designed to help them connect with their difficult emotions and experiences in a flexible way, and improve emotional well-being.

SUMMARY:
The goal of this pilot study is to determine the feasibility, acceptability and impact of a brief behavioral intervention - the "Well-Beans for Caregivers" program, for adult caregivers of individuals with tuberous sclerosis complex (TSC) of any age. The main questions of the study are:

1. Can this innovative, ultra-brief caregiver well-being intervention be delivered feasibly to caregivers via an online modality?
2. How do the caregivers experience the program (acceptability)?
3. Does limited efficacy testing suggest the program has an impact on caregiver's well-being?

DETAILED DESCRIPTION:
The investigators hypothesize that an innovative, ultra-brief caregiver wellbeing intervention developed for caregivers of children with developmental disabilities can be adapted as a universal caregiver wellbeing intervention in tuberous sclerosis complex (TSC), that it can be delivered feasibly in an online modality, and will result in changes in key caregiver wellbeing factors. To test these hypotheses, the researchers will adapt the 3-session 'Well-Beans for Caregivers' program through a participatory method with the TAND consortium (the TAND consortium is an international group of clinical and research professionals as well as family members living with individuals with TSC - TAND stands for TSC-Associated Neuropsychiatric Disorders - see tandconsortium.org). The input from the TAND Consortium will be augmented by members of TSCi (Tuberous Sclerosis International), the global network of TSC non-profit organizations.

For step 2 (pilot intervention), two specialist facilitators and four trainee observers will deliver the 3-session program using ZoomPro, a secure online platform to two groups of 10-12 caregivers. Caregivers are those who provide long-term, day-to-day support and care, and this group includes parents, partners, relatives, or other family members (not paid professional caregivers). These sessions will not be recorded to ensure that participants can join the program without feeling concerned about being recorded. Data collection will use a quasi-experimental pre-post-test design. Eligible and consented participants will therefore complete baseline data as 'pre-test' and then 'post-test' data after the 3-week intervention. Following this, they will complete 3-month and 6-month data collection. Caregiver wellbeing measures will only include open access and freely available measures. The program as well as data collection will be conducted in English.

ELIGIBILITY:
Inclusion Criteria:

* Adult caregiver of an individual with Tuberous Sclerosis Complex (TSC) of any age

Exclusion Criteria:

* Not an adult caregiver of an individual with TSC

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Attendance rates to assess feasibility | At the end of cycle 1, cycle 2 and cycle 3 (each cycle is 7 days)
  Attendance rates at each of the three weekly intervention sessions will be tracked as a measure of feasibility of the intervention program.
Feasibility Feedback Forms for caregivers, facilitators and observers | At the end of cycle 1, cycle 2 and cycle 3 (each cycle is 7 days)
  Caregivers, facilitators and observers will complete bespoke Feasibility Feedback Forms to assess whether the intervention could be implemented as designed.
Acceptability Feedback Forms for caregivers, facilitators and observers | At the end of cycle 1, cycle 2 and cycle 3 (each cycle is 7 days)
  Caregivers, facilitators and observers will complete bespoke Acceptability Feedback Forms to assess their experience and acceptability of the program.

SECONDARY OUTCOMES:
Change in psychological flexibility on the Psy-Flex measure | Change from baseline to immediately post-treatment, and at 3 and 6 months post-treatment
  Changes in scores on the Psy-Flex (Gloster, 2021) will be used to assess changes in caregiver psychological flexibility from before to after treatment. The Psy-Flex consists of 6 items with a minimum score of 6 and a maximum score of 30. Higher scores indicate better psychological flexibility (better outcome).
Change in depression on the Patient Health Questionnaire-9 (PHQ-9) | Change from baseline to immediately post-, and 3 and 6-month post treatment
  Changes in participant levels of depression will be measured via changes in scores on the Patient Health Questionnaire (PHQ-9) from before to after the intervention and at two follow-up intervals. The PHQ consists of 9 items with a minimum score of 0 and a maximum score of 27. Higher scores indicate higher levels of depression.
Change in anxiety on the Generalized Anxiety Disorder-7 Scale (GAD-7) | Change from baseline to immediately post-, and 3 and 6-month post treatment
  Changes in anxiety will be assessed via changes in scores on the Generalized Anxiety Disorder-7 Scale (GAD-7). This is a 7-item scale with a minimum score of 0 and a maximum score of 21. Higher scores indicate higher levels of anxiety.
Change in general wellbeing scores on the World Health Organization Wellbeing Index (WHO-5) | Change from baseline to immediately post-, and 3 and 6-month post treatment
  Changes in general wellbeing will be assessed via changes in scores on the WHO-5 Wellbeing Index (WHO-5). This is a 5-item scale with a minimum score of 0 and a maximum score of 25. Higher scores indicate higher levels of well-being.
Change in resilience as measured on the Brief Resilience Scale | Change from baseline to immediately post-, and 3 and 6-month post treatment
  Changes in resilience will be assessed via changes in scores on the Brief Resilience Scale (BRS). The BRS is a 6-item scale with a minimum score of 6 and a maximum score of 30. Higher scores indicate higher levels of resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Jansen, MD, PhD, Principal Investigator — Vrije Universiteit Brussel; Petrus J de Vries, MD PhD, Principal Investigator — University of Cape Town
Locations (2):
- TSC Alliance, Silver Spring, Maryland, United States
- Tuberous Sclerosis Australia, Beverly Hills, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schlebusch L, Chambers N, Rosenstein D, Erasmus P; WHO CST Team; de Vries PJ. Supporting caregivers of children with developmental disabilities: Findings from a brief caregiver well-being programme in South Africa. Autism. 2024 Jan;28(1):199-214. doi: 10.1177/13623613221133182. Epub 2022 Nov 9. PMID 36352758